CLINICAL TRIAL: NCT00529958
Title: A Randomized Clinical Trial Comparing Three Methods for Anterior Cruciate Ligament Reconstruction: Patellar Tendon, Quadruple Semitendinosus/Gracilis and Double-Bundle Semitendinosus/Gracilis Grafts.
Brief Title: Comparison of Three Methods for Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Workers' Compensation Board, Alberta (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Mohtadi, Clinical Professor and Orthopaedic Surgeon, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB15-1061 (formerly 20966)
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Anterior Cruciate Ligament Rupture; Deficiency of Anterior Cruciate Ligament; Chronic Instability of Knee; Anterior Cruciate Ligament Injury
Keywords: Anterior Cruciate Ligament (ACL) Reconstruction; Patellar Tendon; Hamstring Tendon; Double-Bundle; Autograft
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Bone-Patellar Tendon-Bone Grafting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patellar Tendon (PT) (Active Comparator): ACL reconstruction using a patellar tendon autograft
  Interventions: Procedure: Patellar Tendon
- Hamstring (HT) (Active Comparator): ACL reconstruction using a quadruple-strand semitendinosus/gracilis (hamstring) tendon single-bundle autograft
  Interventions: Procedure: Hamstring Tendon
- Double-Bundle (DB) (Active Comparator): ACL reconstruction using a semitendinosus/gracilis (hamstring) tendon double-bundle autograft
  Interventions: Procedure: Double-Bundle

INTERVENTIONS:
Procedure: Patellar Tendon — Patellar Tendon autograft
  Other Names: Bone-patellar tendon-bone graft; BTPB graft
  Arms: Patellar Tendon (PT)
Procedure: Hamstring Tendon — Quadruple Semitendinosus/Gracilis (Hamstring) Tendon Autograft
  Other Names: Single-bundle hamstring graft; ST/G graft
  Arms: Hamstring (HT)
Procedure: Double-Bundle — Double-Bundle Semitendinosus/Gracilis (Hamstring) Tendon Autograft
  Other Names: Double-bundle ST/G graft
  Arms: Double-Bundle (DB)

SUMMARY:
The purpose of this randomized clinical trial is to determine the difference in quality of life outcome at two years, in patients undergoing an Anterior Cruciate Ligament (ACL) reconstruction procedure with either a patellar tendon, quadruple hamstring tendon or a double-bundle hamstring tendon autograft.

DETAILED DESCRIPTION:
Following an ACL injury, the knee is predisposed to chronic instability, further damage to the meniscal and chondral structures in the knee, osteoarthritis and an impaired quality of life. The successful treatment of an ACL deficient knee aims to preserve the intact meniscus and chondral structures, and to provide a functionally stable knee so that patients can return to pre-injury activities and restore their quality of life. The current standard of care for ACL deficient knees is with a surgical ACL reconstruction procedure. A Cochrane Review was done and demonstrated that the existing literature is controversial. To date, no existing trial has used validated patient-based outcome assessment, accounted for the critical differences between acute and chronic ACL deficiency or used modern techniques to ensure randomization concealment and a sufficient sample size to avoid type II error. The existing information does not define graft failure or re-ruptures, involve long-term follow-up to address osteoarthritis development, nor compare outcomes between single- and double-bundle reconstructive techniques. The current standard includes either a patellar tendon or quadruple semitendinosus/gracilis tendon autograft reconstruction. The newest option is a double-bundle semitendinosus/gracilis graft. This option attempts to restore the complex ACL anatomy by using two separate tendon components to reconstruct the ACL. This study will measure disease-specific quality of life at short- and long-term post-operative intervals (1, 2, 5 and 10 years). Additional secondary outcomes, including the incidence of traumatic re-ruptures and graft failures, will also be compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

A confirmed diagnosis of anterior cruciate ligament deficiency based on all of the following:

* History of a traumatic injury episode
* Physical examination findings of increased anterior translation of the tibia on the femur (Lachman test and/or anterior drawer test)
* A positive pivot shift test
* X-rays showing skeletal maturity (ie: tibial tubercle fused) and no fractures. (NB: Magnetic resonance imaging is not required)
* Age 14-50 years old

Exclusion Criteria:

* Patients with combined ligament deficiencies (Posterior Cruciate, Medial and/or Lateral Collateral deficiency.) (NB: Grade 1 side to side differences (ie. < 5mm) on valgus, varus or posterior stress testing will not be considered exclusions)
* Intra-operative identification of International Cartilage Repair Society (ICRS) Grade 4 chondral lesion of > 1 cm ² [61]
* Previous ligament surgery on the affected or contralateral knees
* Cases involving litigation or Worker's Compensation
* Confirmed connective tissue disorder (ie: Ehlers-Danlos, Marfans)
* X-ray showing that tibial physis is not fused

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2023-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas G Mohtadi, MD MSc FRCSC, Principal Investigator — University of Calgary Sport Medicine Centre
Locations (1):
- University of Calgary Sport Medicine Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohtadi N. Development and validation of the quality of life outcome measure (questionnaire) for chronic anterior cruciate ligament deficiency. Am J Sports Med. 1998 May-Jun;26(3):350-9. doi: 10.1177/03635465980260030201. PMID 9617395
- [Background] Mohtadi NG, Chan DS, Dainty KN, Whelan DB. Patellar tendon versus hamstring tendon autograft for anterior cruciate ligament rupture in adults. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD005960. doi: 10.1002/14651858.CD005960.pub2. PMID 21901700
- [Result] Mohtadi N, Barber R, Chan D, Paolucci EO. Complications and Adverse Events of a Randomized Clinical Trial Comparing 3 Graft Types for ACL Reconstruction. Clin J Sport Med. 2016 May;26(3):182-9. doi: 10.1097/JSM.0000000000000202. PMID 25881568
- [Result] Mohtadi N, Chan D, Barber R, Oddone Paolucci E. A Randomized Clinical Trial Comparing Patellar Tendon, Hamstring Tendon, and Double-Bundle ACL Reconstructions: Patient-Reported and Clinical Outcomes at a Minimal 2-Year Follow-up. Clin J Sport Med. 2015 Jul;25(4):321-31. doi: 10.1097/JSM.0000000000000165. PMID 25514139
- [Result] Mohtadi N, Chan D, Barber R, Paolucci EO. Reruptures, Reinjuries, and Revisions at a Minimum 2-Year Follow-up: A Randomized Clinical Trial Comparing 3 Graft Types for ACL Reconstruction. Clin J Sport Med. 2016 Mar;26(2):96-107. doi: 10.1097/JSM.0000000000000209. PMID 26164058
- [Result] Mohtadi NG, Chan DS. A Randomized Clinical Trial Comparing Patellar Tendon, Hamstring Tendon, and Double-Bundle ACL Reconstructions: Patient-Reported and Clinical Outcomes at 5-Year Follow-up. J Bone Joint Surg Am. 2019 Jun 5;101(11):949-960. doi: 10.2106/JBJS.18.01322. PMID 31169571

RESULTS

PARTICIPANT FLOW:
Period: 2-Year Follow-up
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Started | 110 | 110 (110 randomized to HT, but there was (n=1) cross-over from the DB group) | 110 (110 randomized to DB, but there was (n=1) cross-over to the HT group)
Completed | 106 | 108 (108 HT patients analyzed excludes n=1 cross-over patient (analyzed on intention-to-treat basis).) | 108 (108 DB patients analyzed include 1 cross-over with HT graft (analyzed on intention-to-treat basis).)
Not Completed | 4 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrawal by Subject | 3 | 0 | 0
Period: 5-Year Follow-up
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Started | 106 | 108 (108 HT patients available for 5-year follow-up excludes n=1 cross-over patient from the DB group) | 108 (108 DB patients available for 5-year follow-up includes n=1 cross-over with a single-bundle HT graft)
Completed | 103 | 105 | 107
Not Completed | 3 | 3 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: N=110 patients were randomized to each study group. One cross-over from the DB group received an HT graft, but was analyzed as part of the DB study group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB) | Total
Number analyzed (Participants) | 110 | 110 | 110 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (9.7) | 28.5 (9.9) | 28.3 (9.8) | 28.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 49 | 147
  Male | 63 | 59 | 61 | 183
Chronicity: Acute, Chronic [Count of Participants; unit: Participants]
  Acute | 16 | 16 | 17 | 49
  Chronic | 94 | 94 | 93 | 281
Injured side: Left, Right [Count of Participants; unit: Participants]
  Left | 54 | 63 | 54 | 171
  Right | 56 | 47 | 56 | 159

OUTCOME MEASURES:

1. Primary Outcome: Anterior Cruciate Ligament Quality of Life (ACL-QOL) Outcome
Description: The 32-item patient-reported Anterior Cruciate Ligament Quality-of-Life (ACL-QOL) questionnaire assesses symptoms/physical complaints, work-related, sports/recreational, lifestyle and social/emotional concerns. A higher score on the 0 to 100mm visual analog scale represents better quality of life.
Time Frame: Baseline, 3 and 6 months, 1, 2, and 5 years post-operatively
Population: There were 110 participants randomized to each study group. At 1- and 2-year follow-up, outcome data was not collected for all participants due to loss-to-follow-up, withdrawal or missed study visits.
Measure: Mean (Standard Deviation); unit: Score (0 to 100)
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Score (0 to 100)
  Baseline | 27.0 (13.1) | 29.8 (14.7) | 28.7 (13.7)
  3 Months: number analyzed (Participants) | 108 | 108 | 108
  3 Months | 47.7 (17.2) | 52.6 (19.2) | 50.5 (16.9)
  6 Months: number analyzed (Participants) | 106 | 105 | 109
  6 Months | 61.7 (19.1) | 65.2 (18.4) | 65.5 (17.9)
  1-Year: number analyzed (Participants) | 103 | 107 | 107
  1-Year | 74.5 (18.7) | 75.4 (18.5) | 73.6 (19.2)
  2-Years: number analyzed (Participants) | 106 | 108 | 108
  2-Years | 84.6 (16.6) | 82.5 (17.7) | 82.4 (17.5)
  5-Years: number analyzed (Participants) | 103 | 105 | 107
  5-Years | 82.5 (17.9) | 83.9 (18.2) | 81.1 (19.3)
Statistical Analysis 1: Comparison: Patellar Tendon (PT) vs Hamstring (HT) vs Double-Bundle (DB); All patients were analyzed on an "intention-to-treat" basis using a 5% significance level for all analyses. The ACL-QOL scores for each study group were analyzed using adjusted Bonferroni comparisons and repeated-measures analyses, using a mixed-model analysis of variance for treatment group over time of assessment; Test type: Equivalence — The sample size calculation was based on 88 ACL-deficient patients with surgical intervention and an ACL-QOL score of 74.5 (SD=20.1) at a mean 39-month follow-up, a minimal clinically important difference of 10 points, power=0.80 and p=0.05; p < 0.05, Mixed Models Analysis — A Bonferroni adjustment for multiple comparisons was used in the sample size calculation, resulting in 90 patients per group. With a 20% lost-to-follow-up rate, the final sample size was 108 patients per group for a total of 324 patients

2. Secondary Outcome: Number of Participants With Traumatic ACL Re-ruptures and Atraumatic Graft Failures
Description: * COMPLETE TRAUMATIC RE-RUPTURE - defined as a consequence of an acute traumatic event resulting in a change in static stability since the most recent follow-up visit; determined clinically by a definite loss of end point on Lachman testing, increased anterior translation (>3mm) and a greater than or equal grade 2 pivot shift. Confirmed by MRI or diagnostic arthroscopy.
  * PARTIAL TRAUMATIC TEARS - defined as a consequence of an acute traumatic event resulting in a suspected meniscal injury or graft tear on history, without the clinical characteristics of a "complete traumatic rerupture". Confirmed by MR or diagnostic arthroscopy.
  * TRAUMATIC RE-INJURY - combined total of "complete traumatic re-ruptures" and "partial traumatic tears".
  * ATRAUMATIC GRAFT FAILURES - defined in the absence of an acute traumatic event, with greater than or equal grade 2 pivot shift and/or greater than or equal to 6mm side-to-side difference on the KT arthrometer.
Time Frame: Minimum 2-year Follow-up, 5-Year Follow-up, 10-Year Follow-up
Population: There were 110 participants randomized to each study group. At 5-year follow-up, outcome data was not collected for all participants due to loss-to-follow-up, withdrawal or missed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  Minimum 2-Year Follow-up: No re-injury or failure | 91 | 81 | 79
  Minimum 2-Year Follow-up: Complete Traumatic Re-rupture | 3 | 7 | 7
  Minimum 2-Year Follow-up: Partial Traumatic Tear | 0 | 5 | 4
  Minimum 2-Year Follow-up: Atraumatic Graft Failure | 16 | 17 | 20
  5-Year Follow-up: number analyzed (Participants) | 103 | 105 | 107
  5-Year Follow-up: No re-injury or failure | 92 | 80 | 76
  5-Year Follow-up: Complete Traumatic Re-rupture | 4 | 11 | 11
  5-Year Follow-up: Partial Traumatic Tear | 0 | 5 | 6
  5-Year Follow-up: Atraumatic Graft Failure | 7 | 9 | 14

3. Secondary Outcome: Number of Participants With Each International Knee Documentation Committee (IKDC) Objective Overall Group Grade
Description: IKDC Objective group grades: Normal (A), Nearly Normal (B), Abnormal (C), Severely Abnormal (D) The IKDC Objective Overall Group Grade is determined by the lowest grade assigned to defined objective knee examination measurements, including effusion, passive motion deficit and manual/instrumented ligament examinations (i.e. Lachman, anterior-posterior (AP) translation).
Time Frame: Baseline, 1, 2, 5 years post-operatively
Population: There were 110 participants randomized to each study group. At 1-, 2-, and 5-year follow-up, outcome data was not collected for all participants due to loss-to-follow-up, withdrawal or missed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  Baseline: number analyzed (Participants) | 109 | 109 | 110
  Baseline: Normal (A) | 0 | 0 | 0
  Baseline: Nearly Normal (B) | 1 | 4 | 5
  Baseline: Abnormal (C) | 103 | 101 | 100
  Baseline: Severely Abnormal (D) | 5 | 4 | 5
  1-Year: number analyzed (Participants) | 101 | 104 | 101
  1-Year: Normal (A) | 9 | 9 | 9
  1-Year: Nearly Normal (B) | 79 | 77 | 71
  1-Year: Abnormal (C) | 13 | 18 | 19
  1-Year: Severely Abnormal (D) | 0 | 0 | 2
  2-Years: number analyzed (Participants) | 101 | 104 | 107
  2-Years: Normal (A) | 12 | 12 | 19
  2-Years: Nearly Normal (B) | 65 | 62 | 56
  2-Years: Abnormal (C) | 23 | 28 | 30
  2-Years: Severely Abnormal (D) | 1 | 2 | 2
  5-Years: number analyzed (Participants) | 98 | 99 | 103
  5-Years: Normal (A) | 24 | 18 | 19
  5-Years: Nearly Normal (B) | 61 | 63 | 58
  5-Years: Abnormal (C) | 13 | 18 | 24
  5-Years: Severely Abnormal (D) | 0 | 0 | 2

4. Secondary Outcome: Mean International Knee Documentation Committee (IKDC) Subjective Score
Description: Patient-reported health-related outcome measure with a score between 0 and 100. A higher score represents a better outcome.
Time Frame: Baseline, 3 and 6 months, 1, 2 and 5 years post-operatively
Population: There were 110 participants randomized to each study group. At 1-, 2- and 5-year follow-up, outcome data was not collected for all participants due to loss-to-follow-up, withdrawal or missed study visits.
Measure: Mean (Standard Deviation); unit: score on a scale (out of 100)
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
score on a scale (out of 100)
  Baseline | 50.1 (13.9) | 51.0 (16.2) | 51.5 (14.6)
  3 Months: number analyzed (Participants) | 105 | 108 | 108
  3 Months | 60.2 (12.2) | 65.7 (14.2) | 63.1 (12.1)
  6 Months: number analyzed (Participants) | 105 | 103 | 109
  6 Months | 71.1 (11.1) | 76.1 (13.1) | 75.8 (11.1)
  1-Year: number analyzed (Participants) | 101 | 105 | 107
  1-Year | 79.7 (11.7) | 81.7 (12.6) | 80.0 (11.9)
  2-Years: number analyzed (Participants) | 105 | 107 | 107
  2-Years | 84.6 (13.8) | 85.3 (11.6) | 84.2 (11.8)
  5-Years: number analyzed (Participants) | 103 | 105 | 107
  5-Years | 83.9 (12.9) | 85.2 (13.0) | 84.3 (13.4)

5. Secondary Outcome: Number of Participants With Each Pivot Shift Grade
Description: The Pivot Shift test is a dynamic, passive test to assess the rotational instability of the Anterior Cruciate Ligament in the knee.
  Pivot shift grades include: equal/0 (negative); glide/1; clunk/2; gross/3. A positive grade indicates injury to the Anterior Cruciate Ligament.
Time Frame: Baseline, 3 and 6 months, 1, 2 and 5 years post-operatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  Baseline: Equal | 0 | 1 | 0
  Baseline: Glide (+) | 6 | 6 | 9
  Baseline: Clunk (++) | 103 | 102 | 99
  Baseline: Gross (+++) | 1 | 1 | 2
  3 Months: number analyzed (Participants) | 104 | 106 | 107
  3 Months: Equal | 73 | 60 | 80
  3 Months: Glide (+) | 30 | 45 | 25
  3 Months: Clunk (++) | 1 | 1 | 2
  3 Months: Gross (+++) | 0 | 0 | 0
  6 Months: number analyzed (Participants) | 103 | 103 | 107
  6 Months: Equal | 62 | 53 | 66
  6 Months: Glide (+) | 38 | 45 | 39
  6 Months: Clunk (++) | 3 | 5 | 2
  6 Months: Gross (+++) | 0 | 0 | 0
  1-Year: number analyzed (Participants) | 101 | 106 | 102
  1-Year: Equal | 47 | 46 | 53
  1-Year: Glide (+) | 51 | 48 | 41
  1-Year: Clunk (++) | 3 | 12 | 7
  1-Year: Gross (+++) | 0 | 0 | 1
  2-Years: number analyzed (Participants) | 102 | 104 | 107
  2-Years: Equal | 36 | 28 | 38
  2-Years: Glide (+) | 52 | 57 | 49
  2-Years: Clunk (++) | 14 | 18 | 19
  2-Years: Gross (+++) | 0 | 1 | 1
  5-Years: number analyzed (Participants) | 99 | 99 | 103
  5-Years: Equal | 37 | 29 | 30
  5-Years: Glide (+) | 50 | 54 | 50
  5-Years: Clunk (++) | 12 | 16 | 22
  5-Years: Gross (+++) | 0 | 0 | 1

6. Secondary Outcome: Proportion of Patients With Moderate or Severe Kneeling Pain
Description: Patients kneeled down on the same hard surface (i.e. clinic floor) and self-reported the pain on a scale of: none, mild, moderate or severe. The number of patients reporting moderate or severe kneeling pain were combined in the reported proportions.
Time Frame: Baseline, 2 and 5 years post-operatively
Population: At 2 and 5-year follow-up, outcome data was not collected on all participants due to loss-to-follow-up, withdrawal or missed study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  Baseline: number analyzed (Participants) | 109 | 110 | 110
  Baseline | 29 | 29 | 18
  2 Years: number analyzed (Participants) | 98 | 103 | 104
  2 Years | 17 | 9 | 4
  5 Years: number analyzed (Participants) | 98 | 98 | 101
  5 Years | 10 | 4 | 2

7. Secondary Outcome: Knee Laxity as Measured by the KT Arthrometer
Description: Mean side-to-side differences, as measured using the KT-1000 Arthrometer instrument at 30lbs/134N forces to objectively measure knee laxity.
Time Frame: Baseline, 1 and 2 years post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimetres (side-to-side difference)
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Millimetres (side-to-side difference)
  Baseline | 4.9 (2.3) | 5.0 (2.1) | 5.1 (2.3)
  1-Year: number analyzed (Participants) | 101 | 106 | 102
  1-Year | 1.9 (2.3) | 2.8 (1.8) | 2.8 (2.2)
  2-Years: number analyzed (Participants) | 102 | 104 | 107
  2-Years | 1.9 (2.5) | 3.0 (2.1) | 2.7 (2.4)

8. Secondary Outcome: Mean Tegner Activity Level
Description: Tegner Activity Scale (Values indicate level of activity from inactive (Level 0) to competitive level of activity (Level 10))
Time Frame: Baseline, 6 months, 1 and 2 years post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Activity Level
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Activity Level
  Baseline | 7.7 (1.7) | 7.9 (1.7) | 7.9 (1.6)
  6 Months: number analyzed (Participants) | 105 | 103 | 109
  6 Months | 4.7 (1.6) | 4.8 (1.6) | 5.0 (1.7)
  1 Year: number analyzed (Participants) | 101 | 105 | 107
  1 Year | 6.0 (1.8) | 6.1 (1.9) | 5.9 (2.0)
  2 Years: number analyzed (Participants) | 103 | 107 | 107
  2 Years | 6.5 (1.8) | 6.4 (2.0) | 6.4 (1.9)

9. Secondary Outcome: Return to Pre-injury Tegner Activity Level
Description: Proportion of patients returning to pre-injury levels, as measured by the Tegner Activity Scale (Values indicate level of activity from inactive (Level 0) to competitive level of activity (Level 10)).
Time Frame: 1, 2 and 5 years post-operatively
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  1 Year | 27 | 33 | 28
  2 Years | 44 | 43 | 36
  5 Years | 35 | 41 | 41

10. Secondary Outcome: Cincinnati Occupational Rating Scale
Description: The Cincinnati Occupational Rating Scale assesses the level of work-related activities, including sitting, standing, walking, squatting, climbing, lifting and carrying weighted objects. The score ranges from 0 to 100, with a lower score representing more sedentary work-related activities.
Time Frame: Baseline, 3 and 6 months, 1, 2 and 5 years post-operatively
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (out of 100)
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
score on a scale (out of 100)
  Baseline | 36.6 (19.9) | 35.4 (21.3) | 36.3 (17.7)
  3 Months: number analyzed (Participants) | 105 | 108 | 108
  3 Months | 34.7 (17.2) | 36.1 (22.1) | 36.4 (19.3)
  6 Months: number analyzed (Participants) | 105 | 102 | 109
  6 Months | 35.7 (18.3) | 37.4 (21.6) | 37.0 (20.2)
  1 Year: number analyzed (Participants) | 101 | 105 | 107
  1 Year | 36.7 (17.2) | 38.0 (22.0) | 38.0 (21.5)
  2 Years: number analyzed (Participants) | 104 | 107 | 107
  2 Years | 36.8 (19.4) | 34.4 (22.1) | 38.0 (22.5)
  5 Years: number analyzed (Participants) | 103 | 105 | 107
  5 Years | 35.9 (18.4) | 36.6 (23.8) | 37.8 (24.2)

11. Secondary Outcome: Skin-to-Skin Operative Times
Description: Skin-to-skin operative times (in minutes) for each ACL reconstruction procedure
Time Frame: During surgery
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Minutes | 75.3 (14.7) | 67.8 (14.6) | 88.0 (14.9)

12. Secondary Outcome: Radiographic (X-ray) Changes
Description: The analysis for the radiographic assessment data is currently ongoing, to provide a comparison of baseline, 2- and 5-year post-operative x-rays.
Time Frame: Baseline, 2 and 5 years post-operatively
Reporting Status: Not Posted, anticipated posting 2025-03

13. Other Pre Specified Outcome: Complications of the Surgical Procedure (See Adverse Events Section for Results of This Outcome)
Description: All complications/adverse events that occurred within the first two-years post-operatively.
  See Adverse Events section for results of this outcome.
Time Frame: 2 years post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
Number analyzed (Participants) | 110 | 110 | 110
Participants
  Deep wound infection | 1 | 0 | 0
  Superficial wound infection | 0 | 2 | 2
  Chondral lesion | 1 | 0 | 1
  Failed meniscal repair | 2 | 6 | 4
  Stiffness | 4 | 2 | 3
  Hamstring injury | 1 | 6 | 12
  Tibial periostitis | 1 | 2 | 4
  Stitch abscess | 2 | 1 | 0
  Cellulitis | 0 | 0 | 3
  Meniscal cyst | 1 | 0 | 0
  Patellar tendinopathy | 1 | 0 | 0
  Persistent effusion / inflammation | 1 | 2 | 5
  Sensory nerve problems | 4 | 1 | 3
  Wound dehiscence | 1 | 0 | 1
  Hardware issues | 0 | 0 | 0
  Massive pulmonary embolism | 0 | 0 | 1
  Deep vein thrombosis | 0 | 0 | 1
  Septic arthritis | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Two years post-operatively.
Description: Patient-reported adverse events by phone, email or at regularly scheduled follow-up visits. Unexpected/unusual problems with the patient's knee were assessed in clinic, diagnosed and managed accordingly. Patients presenting with emergent concerns were initially seen in the hospital emergency department. All patients experiencing an adverse event/complication were followed (by phone, email, regularly scheduled or additional visits) until the issue was completely resolved or appropriately managed.
Arm/Group | Patellar Tendon (PT) | Hamstring (HT) | Double-Bundle (DB)
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110 | 1/110 | 2/110
Other Adverse Events (participants affected / at risk) | 20/110 | 22/110 | 38/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patellar Tendon (PT) (N=110) | Hamstring (HT) (N=110) | Double-Bundle (DB) (N=110)
Septic Arthritis (Infections and infestations) | 0 | 1 | 0 — Detected 1 month post-operatively; treated with arthroscopic washout, intravenous antibiotics and successful preservation of the graft. Coagulase-negative Staphylococcus was the identified organism. Complete resolution.
Massive Pulmonary Embolism (Blood and lymphatic system disorders) | 0 | 0 | 1 — Identified at 2 weeks post-operatively; treated successfully with anticoagulation and an IVC filter with no long-term sequelae. Complete resolution.
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 — Identified 18 days post-operatively; treated successfully with anticoagulant therapy with no clinical sequelae.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patellar Tendon (PT) (N=110) | Hamstring (HT) (N=110) | Double-Bundle (DB) (N=110)
Failed Meniscal Repair (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4 — Requiring repeat surgery for medial meniscal tears. There were no lateral meniscal tears.
Stiffness (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 — Intra-articular scarring requiring repeat surgery, caused by generalized arthrofibrosis (1), Cyclops lesions (4), or graft hypertrophy causing impingement (4).
Hamstring Injury (Musculoskeletal and connective tissue disorders) | 1 | 6 | 12 — Hamstring injuries on the ipsilateral side, include hamstring strain (18 patients) and a hamstring tear (1 patient with a patellar tendon graft; tear due to a major traumatic event while wakeboarding).
Tibial Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 — Diagnosed as pain, swelling, redness and tenderness isolated to the medial tibial surface, distinct from pain in the knee. All presented within 2 weeks post-operatively; all successfully treated with nonsteroidal anti-inflammatory drugs (NSAIDS)
Deep Wound Infection (Infections and infestations) | 1 | 0 | 0 — Treated successfully with IV and oral antibiotics
Superficial Wound Infection (Infections and infestations) | 0 | 2 | 2 — Successfully treated with oral antibiotics.
Sensory Nerve Problems (Nervous system disorders) | 4 | 1 | 3 — Related to graft harvest/portal incisions (5 patients) or as a result of medial meniscal repair (3 patients); treated with topical NSAIDs cream and corticosteroid injections. All problems were resolved except one resulting in long-term dysesthesia.
Stitch Abscess (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Cellulitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Meniscal Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Patellar Tendinopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Chondral Lesion (Metabolism and nutrition disorders) | 1 | 0 | 1 — Requiring surgery.
Persistent Effusion/Inflammation (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Hardware Issues (Surgical and medical procedures) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No